CLINICAL TRIAL: NCT07294144
Title: A Study to Evaluate the Biological Effect of Tofersen in Adults With Amyotrophic Lateral Sclerosis Without Mutations in SOD1
Brief Title: Tofersen in Non-SOD1 ALS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Timothy M. Miller, MD, PhD, David Clayson Professor of Neurology, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US-TOF-12361
Record Dates: First submitted 2025-12-15; First posted 2025-12-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
Keywords: als; amyotrophic lateral sclerosis; tofersen; qalsody
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — tofersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tofersen (Experimental)
  Interventions: Drug: Tofersen

INTERVENTIONS:
Drug: Tofersen — Tofersen 100 mg administered intrathecally.

SUMMARY:
The goal of this clinical trial is to evaluate whether tofersen is safe and effective in adults with non-SOD1 ALS. Tofersen is currently approved by the U.S. Food and Drug Administration to treat SOD1-ALS. The main questions it aims to answer are:

* Does tofersen lower the levels of neurofilament light chain (NfL) in the blood and CSF of adult participants with non-SOD1 ALS?
* Is tofersen safe and tolerable for adult participants with non-SOD1 ALS?
* Does tofersen affect other measurements such as clinical outcomes and quality-of-life measures in participants with non-SOD1 ALS?

Participants will :

* Receive 100mg tofersen via lumbar puncture for 24 weeks. The doses are at the following time points: Weeks 0, 2, 4, 8, 12, 16, 20, and 24.
* Complete 2 follow-up visits following the end of the dosing period at Weeks 28 and 32.
* Complete a variety of questionnaires and outcome measurements such as strength and breathing testing.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use PHI in accordance with national and local participant privacy regulations.
* Aged 18 years or older at the time of informed consent.
* Confirmed diagnosis of ALS.
* Time since onset of weakness due to ALS ≤ 24 months at the time of the screening visit.
* Prior confirmed genetic testing negative for SOD1 and FUS mutations. Participants with mutations in genes other than SOD1 and FUS may be enrolled at the discretion of the Site Investigator.
* SVC ≥ 50% of predicted value as adjusted for sex, age, and height (from the sitting position).
* Medically able to undergo the study procedures and to adhere to the visit schedule at the time of study entry, as determined by the Investigator.
* All participants must agree to practice effective contraception during the study and be willing and able to continue contraception for 5 months after their last dose of study treatment.
* If taking riluzole, participant must be on a stable dose for ≥ 30 days prior to Day 1 and expected to remain at that dose until the final study visit.
* If taking edaravone, participant must have initiated edaravone ≥ 60 days (2 treatment cycles) prior to Day 1 and expected to remain at that dose until the final study visit, unless the Investigator determines that edaravone should be discontinued for medical reasons, in which case it may not be restarted during the study.

Exclusion Criteria:

* Treatment with another investigational drug (including investigational drugs for ALS through compassionate use or expanded access programs), biological agent, or device within 1 month or 5 half-lives of study agent, whichever is longer. Specifically, no prior treatment with small interfering RNA, stem cell therapy, or gene therapy is allowed.
* Current enrollment in any other interventional study.
* History of drug abuse or alcoholism within ≤ 6 months of study enrollment that would limit participation in the study, as determined by the Investigator.
* Presence of an untreated or inadequately treated active infection requiring systemic antiviral or antimicrobial therapy at any time during the screening period.
* Ongoing medical condition (e.g., wasting or cachexia, severe anemia) that according to the Investigator would interfere with the conduct or assessments of the study.
* History of confounding neuromuscular or neurological disorder that is expected to have a progressive (i.e., worsening) course during the study, and/or is expected to be associated with elevations in neurofilament, in the opinion of the Investigator.
* Female participants who are pregnant or currently breastfeeding.
* Significant cognitive impairment, clinical dementia, or unstable psychiatric illness, including psychosis, suicidal ideation, suicide attempt, or untreated major depression ≤ 90 days, as determined by the Investigator.
* History of allergies to a broad range of anesthetics.
* Tracheostomy.
* Presence of risk for increased or uncontrolled bleeding and/or risk of bleeding that is not managed optimally could place a participant at an increased risk for intraoperative or postoperative bleeding. These could include, but are not limited to, anatomical factors at or near the LP site (e.g., vascular abnormalities, neoplasms, or other abnormalities) and underlying disorders of the coagulation cascade, platelet function, or platelet count (e.g., hemophilia, Von Willebrand's disease, liver disease).
* Anticipated need, in the opinion of the Investigator, for administration of any antiplatelet or anticoagulant medication that cannot be safely held before and/or after an LP procedure according to local or institutional guidelines and/or Investigator determination.
* Presence of an implanted shunt for the drainage of CSF or an implanted CNS catheter.
* Clinically significant abnormalities in hematology or clinical chemistry parameters, as determined by the Investigator, which would render the participant unsuitable for enrollment.
* Inability to comply with study requirements.
* Other unspecified reasons that, in the opinion of the Investigator, make the participant unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with ≥30% reduction in plasma NfL | From Baseline to Week 28

SECONDARY OUTCOMES:
Proportion of participants with ≥ 30% reduction in CSF NfL | From Baseline to Week 28
Change in plasma and CSF NfL levels | From Baseline to Week 28
Incidence of adverse events and serious adverse events | From Baseline through study completion, an average of 8 months

OTHER OUTCOMES:
Changes in CSF SOD1 | From Baseline to Week 28
Change in ALS Functional Rating Scale - Revised (ALSFRS-R) | From Baseline to Week 28
  The ALSFRS-R measures 4 functional domains, including respiratory, bulbar function, gross motor skills, and fine motor skills. There are 12 questions, each scored from 0 to 4, for a total possible score of 48, with higher scores representing better function.
Change in Slow Vital Capacity (SVC) | From Baseline to Week 28
  Vital capacity will be measured by means of a slow vital capacity test, performed following a standardized protocol established by the Northeast ALS Consortium.
Change in Handheld Dynamometry (HHD) | From Baseline to Week 28
  Quantitative muscle strength will be evaluated using HHD of multiple muscles using standard participant positioning.
Change in Rasch Overall ALS Disability Scale (ROADS) | From Baseline to Week 28
  The Rasch-built Overall ALS Disability Scale (ROADS) is a patient-reported outcome measure that assesses 28 items, each scored 0-2, and then provides a normed total score from 0-146 to capture overall disability level in a linearly-weighted manner, meaning that a 1-point change on the normed ROADS score represents a quantifiable and consistent measurement of disability, and a 2-point change reflects twice the amount of disability.
Change in Motor Functional Independence Measure (FIM) | From Baseline to Week 28
  The Motor Functional Independence Measure (FIM) consists of 13 items assessing motor function scored 0-7, for a maximum score of 91, which indicates the highest level of function.
Change in EuroQol 5-dimension, 5-level scale (EQ-5D-5L) | From Baseline to Week 28
  The EuroQol Five Dimension (EQ-5D-5L) is a standardized generic measure of health status and consists of 2 sections. The first section comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D-5L measures the dimensions on a 5-point scale: no problems, slight problems, moderate problems, severe problems, and extreme problems. The second section comprises the visual analogue scale that records the respondent's self-rated health on a vertical scale ranging from 0 to 100 where the endpoints are labelled "best imaginable health state" and "worst imaginable health state."
Change in ALS Assessment Questionnaire, 5-item scale (ALSAQ-5) | From Baseline to Week 28
  The ALSAQ-5 is a disease-specific self-reported health status questionnaire. The ALSAQ-5 contains 5 questions, each corresponding to 1 of the following 5 health-related dimensions: physical mobility, activities of daily living, eating and drinking abilities, communication, and emotional functioning. The questions are followed by 5 responses with the raw scores ranging from 0 = Never to 4 = Always or cannot do at all. The ALSAQ-5 total score ranges from 0 to 100 with a lower score representing a better health-related status.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University ALS Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No